CLINICAL TRIAL: NCT06052631
Title: Microneurographic Assessment of Peripheral Nerves in Healthy Volunteers and Individuals With Sensory Dysfunction Caused by Inherited Mutations in the PIEZO2 Gene
Status: Recruiting | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001678; 001678-AT
Record Dates: First submitted 2023-09-22; First posted 2023-09-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-29

CONDITIONS: PIEZO2-Deficiency Syndrome
Keywords: Sensation; TOUCH; Proprioception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy participants
- PIEZO2 Deficiency Syndrome (PDS): Participants with a diagnosis of PIEZO2 Deficiency Syndrome; an inherited mutation in the PIEZO2 gene

SUMMARY:
Background:

PIEZO2 Deficiency Syndrome (PDS) is a genetic disorder that affects a person s ability to feel touches and pain. Researchers want to know more about how PDS changes nerve function.

Objective:

To compare nerve function in people with PDS to that in people without PDS.

Eligibility:

People aged 18 years and older with PDS enrolled in protocol 16-AT-0077. Healthy volunteers are also needed.

Design:

Participants will have at least 1 clinic visit. They will undergo a test that measures activity in the nerves.

For the test:

Participants will place their arm or leg in a comfortable position.

Ultrasound will be used to locate nerves. A smooth wand will be slid over the skin to capture images of the structures below.

Two thin needles will be inserted through the skin. These needles are much smaller than the kind used to draw blood.

The needles will record nerve activity as different sensations are applied to the skin. These include mild electrical pulses; heat and cold; bending of the knee or elbow; vibration; air puffs; pulling a hair; and tapping, stroking (brushing), stretching, pinching, and pushing on the skin at different levels of force.

Each test takes 5 to 10 minutes. Participants will describe the sensations they feel.

Participants may opt for an additional test that measures how nerves respond after heat pulses are used to create mild redness on the skin.

Researchers would like at least 2 tests from each person. Participants may return for up to 3 additional visits, if desired, to complete all the testing.

DETAILED DESCRIPTION:
Study Description:

The study aims to characterize peripheral nerve function and physiology in healthy participants and participants with inherited mutations in the PIEZO2 gene (otherwise known as PIEZO2- Deficiency Syndrome [PDS]). PIEZO2 encodes a stretch-gated ion channel whose function has been shown to be essential for aspects of gentle touch sensation, vibration detection, mechanical allodynia and proprioception in humans. The physiological effects of PIEZO2 mutations on sensory neurons in humans are unknown. The study will improve our understanding of the molecular mechanisms for touch and mechanical pain sensation and determine if the peripheral neurons remain otherwise healthy in the absence of a functioning PIEZO2 channel.

Objectives:

Primary Objective:

To determine whether peripheral neurons have a blunted response to gentle mechanical stimulation (e.g., soft brushing) in PDS patients compared to healthy participants using direct electrical recording from peripheral nerves.

Secondary Objectives:

To examine the physiological properties of different types of mechanically sensitive sensory neurons in response to innocuous and noxious stimuli in PDS patients and healthy participants. We expect the loss of PIEZO2 to have greater impact on the responsiveness of certain types mechano-receptor subtypes over others.

Endpoints:

Primary Endpoint:

Our primary endpoint is evidence of reduced responsiveness (i.e., firing rate [Hz]) of peripheral neurons to gentle mechanical (brushing) stimulation in PDS patients compared to controls. We expect a reduction of at least 50% in firing rate (Hz).

Secondary Endpoints:

Our secondary endpoint is the emergence of a differential effect of the loss of PIEZO2 on mechanoreceptor subclasses. Mechanoreceptor subclasses will be identified using established criteria (e.g., stimulus sensitivity, receptive field size, spike morphology and axon conduction velocity). The effect of the loss of PIEZO2 on the responsiveness of single-unit subclasses will be quantified by firing rate measures on single-unit data. In addition, the percept evoked to intraneural electrical stimulation of single-unit subclasses will be noted.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

All Participants

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years and over.
* The ability to provide written informed consent.
* Enrolled in 16-AT-0077, "Clinical and Scientific Assessment of Pain and Painful Disorders".

PDS Patients

-Clinical and genetic diagnosis of PIEZO2-LOF.

Healthy participants

-In good general health as evidenced by medical evaluation under 16-AT-0077.

EXCLUSION CRITERIA:

All Participants:

* Difficulties with communication that make subjective innocuous and pain assessments impossible or unreliable.
* Unable to comply with study procedures or visits.
* Has a dermatological condition that might influence cutaneous sensitivity.
* Congenital limb deficiency or amputation of any limb.
* Prior history of syncope.
* Peripheral neuropathy or current chronic pain condition or has had chronic pain in the past year (painful condition lasting more than six months), including ongoing treatment with medications for neuropathic pain (e.g. gabapentin, tricyclic antidepressants, pregabalin, tramadol).
* Has a major medical condition, such as kidney, liver, cardiovascular, autonomic, pulmonary, or neurological problems (e.g., epilepsy) or a chronic systemic disease (e.g., diabetes), or Raynaud's Disease.
* Current and untreated diagnosis of depression, post-traumatic stress, syndrome, bipolar disorder, psychosis, anxiety or panic disorder, alcohol or substance use disorders.
* Pregnant (verbal confirmation) or breastfeeding.
* Are participating in other ongoing research protocols involving interventions that would interfere with somatosensation.
* Employees or staff that work at NCCIH.
* Adults who are unable to provide their own consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be screened and selected from an existing NCCIH protocol, 16-AT-0077. PDS participants will be referred to 16-AT-0077 for screening from an existing NINDS protocol, 12-N-0095.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Firing rate (Hz) in response to fast and slow brushing. | At each visit (max of 4 visits) during microneurography procedure.
  PDS patients have major deficits in touch detection. Therefore, we predict the response (firing rate) to gentle brush stimuli to be reduced by at least 50% (compared to healthy controls), corresponding to decreased sensitivity to mechanical stimuli. The neural measure of firing rate (Hz) captures both the magnitude of the response and its temporal pattern and has been shown to reliably distinguish between normal and pathological responses and the effects of pharmacological manipulations.

SECONDARY OUTCOMES:
Firing rate (Hz) in response to other sensory modalities, e.g., thermal, and other mechanical stimuli. | At each visit (max of 4 visits) during microneurography procedure.
  Our secondary endpoint is the emergence of a differential effect of the loss of PIEZO2 on mechanoreceptor subclasses. Mechanoreceptor subclasses will be identified using established criteria (e.g., stimulus sensitivity, receptive field size, spike morphology and axon conduction velocity). The effect of the loss of PIEZO2 on the responsiveness of single-unit subclasses will be quantified by firing rate measures on single-unit data. In addition, the percept evoked to intraneural electrical stimulation of single-unit subclasses will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Backonja, M.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesler AT, Szczot M, Bharucha-Goebel D, Ceko M, Donkervoort S, Laubacher C, Hayes LH, Alter K, Zampieri C, Stanley C, Innes AM, Mah JK, Grosmann CM, Bradley N, Nguyen D, Foley AR, Le Pichon CE, Bonnemann CG. The Role of PIEZO2 in Human Mechanosensation. N Engl J Med. 2016 Oct 6;375(14):1355-1364. doi: 10.1056/NEJMoa1602812. Epub 2016 Sep 21. PMID 27653382
- [Background] Case LK, Liljencrantz J, Madian N, Necaise A, Tubbs J, McCall M, Bradson ML, Szczot M, Pitcher MH, Ghitani N, Frangos E, Cole J, Bharucha-Goebel D, Saade D, Ogata T, Donkervoort S, Foley AR, Bonnemann CG, Olausson H, Bushnell MC, Chesler AT. Innocuous pressure sensation requires A-type afferents but not functional RhoIotaEpsilonZetaOmicron2 channels in humans. Nat Commun. 2021 Jan 28;12(1):657. doi: 10.1038/s41467-021-20939-5. PMID 33510158
- [Background] Nagi SS, Marshall AG, Makdani A, Jarocka E, Liljencrantz J, Ridderstrom M, Shaikh S, O'Neill F, Saade D, Donkervoort S, Foley AR, Minde J, Trulsson M, Cole J, Bonnemann CG, Chesler AT, Bushnell MC, McGlone F, Olausson H. An ultrafast system for signaling mechanical pain in human skin. Sci Adv. 2019 Jul 3;5(7):eaaw1297. doi: 10.1126/sciadv.aaw1297. eCollection 2019 Jul. PMID 31281886
- [Background] Curry TB, Charkoudian N. The use of real-time ultrasound in microneurography. Auton Neurosci. 2011 Jul 5;162(1-2):89-93. doi: 10.1016/j.autneu.2011.03.007. Epub 2011 Apr 22. PMID 21514900
- [Background] Delle Vedove A, Storbeck M, Heller R, Holker I, Hebbar M, Shukla A, Magnusson O, Cirak S, Girisha KM, O'Driscoll M, Loeys B, Wirth B. Biallelic Loss of Proprioception-Related PIEZO2 Causes Muscular Atrophy with Perinatal Respiratory Distress, Arthrogryposis, and Scoliosis. Am J Hum Genet. 2016 Nov 3;99(5):1206-1216. doi: 10.1016/j.ajhg.2016.09.019. Epub 2016 Oct 27. PMID 27843126
- [Background] Dunham JP, Sales AC, Pickering AE. Ultrasound-guided, open-source microneurography: Approaches to improve recordings from peripheral nerves in man. Clin Neurophysiol. 2018 Nov;129(11):2475-2481. doi: 10.1016/j.clinph.2018.07.011. Epub 2018 Jul 29. PMID 30107982
- [Background] Eckberg DL, Wallin BG, Fagius J, Lundberg L, Torebjork HE. Prospective study of symptoms after human microneurography. Acta Physiol Scand. 1989 Dec;137(4):567-9. doi: 10.1111/j.1748-1716.1989.tb08804.x. No abstract available. PMID 2690582
- [Background] Edin BB, Abbs JH. Finger movement responses of cutaneous mechanoreceptors in the dorsal skin of the human hand. J Neurophysiol. 1991 Mar;65(3):657-70. doi: 10.1152/jn.1991.65.3.657. PMID 2051199
- [Background] Gandevia SC, Hales JP. The methodology and scope of human microneurography. J Neurosci Methods. 1997 Jun 27;74(2):123-36. doi: 10.1016/s0165-0270(97)02243-7. PMID 9219882
- [Background] Guo YR, MacKinnon R. Structure-based membrane dome mechanism for Piezo mechanosensitivity. Elife. 2017 Dec 12;6:e33660. doi: 10.7554/eLife.33660. PMID 29231809
- [Background] Hagbarth KE. Exteroceptive, proprioceptive, and sympathetic activity recorded with microelectrodes from human peripheral nerves. Mayo Clin Proc. 1979 Jun;54(6):353-65. PMID 156292
- [Background] Haliloglu G, Becker K, Temucin C, Talim B, Kucuksahin N, Pergande M, Motameny S, Nurnberg P, Aydingoz U, Topaloglu H, Cirak S. Recessive PIEZO2 stop mutation causes distal arthrogryposis with distal muscle weakness, scoliosis and proprioception defects. J Hum Genet. 2017 Apr;62(4):497-501. doi: 10.1038/jhg.2016.153. Epub 2016 Dec 15. PMID 27974811
- [Background] Hissen SL, Fu Q. Neural control of blood pressure during pregnancy in humans. Clin Auton Res. 2020 Oct;30(5):423-431. doi: 10.1007/s10286-020-00703-3. Epub 2020 Jun 20. PMID 32564162
- [Background] Le Pichon CE, Chesler AT. The functional and anatomical dissection of somatosensory subpopulations using mouse genetics. Front Neuroanat. 2014 Apr 22;8:21. doi: 10.3389/fnana.2014.00021. eCollection 2014. PMID 24795573
- [Background] Lewis AH, Grandl J. Inactivation Kinetics and Mechanical Gating of Piezo1 Ion Channels Depend on Subdomains within the Cap. Cell Rep. 2020 Jan 21;30(3):870-880.e2. doi: 10.1016/j.celrep.2019.12.040. PMID 31968259
- [Background] Lin YC, Guo YR, Miyagi A, Levring J, MacKinnon R, Scheuring S. Force-induced conformational changes in PIEZO1. Nature. 2019 Sep;573(7773):230-234. doi: 10.1038/s41586-019-1499-2. Epub 2019 Aug 21. PMID 31435018
- [Background] Loken LS, Wessberg J, Morrison I, McGlone F, Olausson H. Coding of pleasant touch by unmyelinated afferents in humans. Nat Neurosci. 2009 May;12(5):547-8. doi: 10.1038/nn.2312. Epub 2009 Apr 12. PMID 19363489
- [Background] Macefield VG, Norcliffe-Kaufmann L, Gutierrez J, Axelrod FB, Kaufmann H. Can loss of muscle spindle afferents explain the ataxic gait in Riley-Day syndrome? Brain. 2011 Nov;134(Pt 11):3198-208. doi: 10.1093/brain/awr168. PMID 22075519
- [Background] Mahmud AA, Nahid NA, Nassif C, Sayeed MS, Ahmed MU, Parveen M, Khalil MI, Islam MM, Nahar Z, Rypens F, Hamdan FF, Rouleau GA, Hasnat A, Michaud JL. Loss of the proprioception and touch sensation channel PIEZO2 in siblings with a progressive form of contractures. Clin Genet. 2017 Mar;91(3):470-475. doi: 10.1111/cge.12850. Epub 2016 Sep 16. PMID 27607563
- [Background] Meah VL, Busch SA, Jones KE, Davenport MH, Steinback CD. A review of acute responses, after-effects and chronic complications related to microneurography. Clin Neurophysiol. 2019 Oct;130(10):1781-1788. doi: 10.1016/j.clinph.2019.06.228. Epub 2019 Jul 15. PMID 31401486
- [Background] Moritz AR, Henriques FC. Studies of Thermal Injury: II. The Relative Importance of Time and Surface Temperature in the Causation of Cutaneous Burns. Am J Pathol. 1947 Sep;23(5):695-720. No abstract available. PMID 19970955
- [Background] Nguyen MQ, Wu Y, Bonilla LS, von Buchholtz LJ, Ryba NJP. Diversity amongst trigeminal neurons revealed by high throughput single cell sequencing. PLoS One. 2017 Sep 28;12(9):e0185543. doi: 10.1371/journal.pone.0185543. eCollection 2017. PMID 28957441
- [Background] Nickolls AR, Lee MM, Espinoza DF, Szczot M, Lam RM, Wang Q, Beers J, Zou J, Nguyen MQ, Solinski HJ, AlJanahi AA, Johnson KR, Ward ME, Chesler AT, Bonnemann CG. Transcriptional Programming of Human Mechanosensory Neuron Subtypes from Pluripotent Stem Cells. Cell Rep. 2020 Jan 21;30(3):932-946.e7. doi: 10.1016/j.celrep.2019.12.062. PMID 31968264
- [Background] Pedersen JL, Kehlet H. Hyperalgesia in a human model of acute inflammatory pain: a methodological study. Pain. 1998 Feb;74(2-3):139-51. doi: 10.1016/s0304-3959(97)00160-7. PMID 9520228
- [Background] Serra J, Duan WR, Locke C, Sola R, Liu W, Nothaft W. Effects of a T-type calcium channel blocker, ABT-639, on spontaneous activity in C-nociceptors in patients with painful diabetic neuropathy: a randomized controlled trial. Pain. 2015 Nov;156(11):2175-2183. doi: 10.1097/j.pain.0000000000000249. PMID 26035253
- [Background] Sharma N, Flaherty K, Lezgiyeva K, Wagner DE, Klein AM, Ginty DD. The emergence of transcriptional identity in somatosensory neurons. Nature. 2020 Jan;577(7790):392-398. doi: 10.1038/s41586-019-1900-1. Epub 2020 Jan 8. PMID 31915380
- [Background] Shy ME, Frohman EM, So YT, Arezzo JC, Cornblath DR, Giuliani MJ, Kincaid JC, Ochoa JL, Parry GJ, Weimer LH; Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Quantitative sensory testing: report of the Therapeutics and Technology Assessment Subcommittee of the American Academy of Neurology. Neurology. 2003 Mar 25;60(6):898-904. doi: 10.1212/01.wnl.0000058546.16985.11. PMID 12654951
- [Background] Szczot M, Liljencrantz J, Ghitani N, Barik A, Lam R, Thompson JH, Bharucha-Goebel D, Saade D, Necaise A, Donkervoort S, Foley AR, Gordon T, Case L, Bushnell MC, Bonnemann CG, Chesler AT. PIEZO2 mediates injury-induced tactile pain in mice and humans. Sci Transl Med. 2018 Oct 10;10(462):eaat9892. doi: 10.1126/scitranslmed.aat9892. PMID 30305456
- [Background] Lemmel EM, Brackertz D, Franke M, Gaus W, Hartl PW, Machalke K, Mielke H, Obert HJ, Peter HH, Sieper J, et al. Results of a multicenter placebo-controlled double-blind randomized phase III clinical study of treatment of rheumatoid arthritis with recombinant interferon-gamma. Rheumatol Int. 1988;8(2):87-93. doi: 10.1007/BF00271840. PMID 3135572
- [Background] Vallbo AB. Microneurography: how it started and how it works. J Neurophysiol. 2018 Sep 1;120(3):1415-1427. doi: 10.1152/jn.00933.2017. Epub 2018 Jun 20. PMID 29924706
- [Background] Vallbo AB, Olausson H, Wessberg J, Kakuda N. Receptive field characteristics of tactile units with myelinated afferents in hairy skin of human subjects. J Physiol. 1995 Mar 15;483 ( Pt 3)(Pt 3):783-95. doi: 10.1113/jphysiol.1995.sp020622. PMID 7776258
- [Background] von Buchholtz LJ, Ghitani N, Lam RM, Licholai JA, Chesler AT, Ryba NJP. Decoding Cellular Mechanisms for Mechanosensory Discrimination. Neuron. 2021 Jan 20;109(2):285-298.e5. doi: 10.1016/j.neuron.2020.10.028. Epub 2020 Nov 12. PMID 33186546
- [Background] Wang Y, Chi S, Guo H, Li G, Wang L, Zhao Q, Rao Y, Zu L, He W, Xiao B. A lever-like transduction pathway for long-distance chemical- and mechano-gating of the mechanosensitive Piezo1 channel. Nat Commun. 2018 Apr 3;9(1):1300. doi: 10.1038/s41467-018-03570-9. PMID 29610524
- [Background] Zhao Q, Zhou H, Chi S, Wang Y, Wang J, Geng J, Wu K, Liu W, Zhang T, Dong MQ, Wang J, Li X, Xiao B. Structure and mechanogating mechanism of the Piezo1 channel. Nature. 2018 Feb 22;554(7693):487-492. doi: 10.1038/nature25743. Epub 2018 Jan 22. PMID 29469092
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001678-AT.html